CLINICAL TRIAL: NCT02784158
Title: An Expanded Access Study of Brigatinib for Patients With ALK-positive Advanced Non-Small Cell Lung Cancer
Status: No longer available | Type: Expanded Access
Sponsor: Ariad Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Other Study IDs: AP26113-16-901
Record Dates: First submitted 2016-05-24; First posted 2016-05-26 (Estimated); Last update posted 2018-02-06 (Actual); Status verified 2018-02

CONDITIONS: Non-small Cell Lung Cancer; Lung Cancer; Advanced Malignancies; Carcinoma
Keywords: Non-small cell lung cancer; Non-small cell lung carcinoma; Epithelial lung cancer; Squamous cell carcinoma; Large cell carcinoma; Adenocarcinoma; Anaplastic lymphoma kinase (ALK); Carcinoma; Advanced Cancers; Brigatinib; AP26113
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms; Carcinoma; Carcinoma, Squamous Cell; Carcinoma, Large Cell; Adenocarcinoma | interventions — brigatinib

INTERVENTIONS:
Drug: Brigatinib — Brigatinib will be administered orally to eligible patients with locally advanced or metastatic ALK+ NSCLC who are resistant or intolerant to a prior ALK inhibitor at a dose of 180 mg QD with a 7 day lead-in at 90 mg QD, continuously, with or without food.
  Other Names: AP26113

SUMMARY:
The purpose of this study is to provide brigatinib for those patients with locally advanced and/or metastatic patients with ALK+ NSCLC on an expanded access basis due to their inability to meet eligibility criteria for on-going recruiting trials, inability to participate in other clinical trials (e.g., poor performance status, lack of geographic proximity), or because other medical interventions are not considered appropriate or acceptable.

ELIGIBILITY:
Inclusion Criteria:

1. Have histologically or cytologically confirmed locally advanced or metastatic NSCLC that is determined to have an ALK-rearrangement detected according to local standard procedure.
2. Resistant to or intolerant of at least 1 prior ALK TKI.
3. Recovered from toxicities related to prior anticancer therapy to NCI CTCAE, v4.0) grade ≤2.
4. Are a male or female patient ≥18 years old.
5. Have adequate organ and hematologic function, as defined by the study protocol.
6. Have Eastern Cooperative Oncology Group (ECOG) performance status ≤2.
7. Have normal QT interval on screening electrocardiogram (ECG) evaluation, defined as QT interval corrected (Fridericia) (QTcF) of ≤450 ms in males or ≤470 ms in females.
8. For female patients of childbearing potential, a negative pregnancy test must be documented prior to enrollment (<7 days prior to the first dose).
9. Female and male patients who are fertile must agree to use a highly effective form of contraception as defined by the study protocol.
10. Must provide a signed and dated informed consent indicating that the patient has been informed of all pertinent aspects of the study, including the potential risks, and is willingly participating.

Exclusion Criteria:

1. Received an ALK TKI within 10 days prior to the first dose of brigatinib.
2. Received cytotoxic chemotherapy, investigational agents, or radiation within 14 days, except stereotactic radiosurgery (SRS) or stereotactic body radiosurgery.
3. Received prior brigatinib therapy.
4. Received monoclonal antibodies within 30 days of the first dose of brigatinib.
5. Had major surgery within 30 days of the first dose of brigatinib.
6. Have current spinal cord compression.
7. Have significant, uncontrolled, or active cardiovascular disease within 6 months prior to first dose, as defined by the study protocol.
8. Have a history or the presence of pulmonary interstitial disease, drug-related pneumonitis, or radiation pneumonitis.
9. Have a known or suspected hypersensitivity to brigatinib or its excipients.
10. Have any condition or illness that, in the opinion of the investigator, would compromise patient safety.
11. Are pregnant or breastfeeding.
12. Are eligible for and have reasonable access to participate in another ongoing brigatinib clinical study.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - UC San Diego Moores Cancer Center (Site 099), La Jolla, California
  - UCI Medical Center-Chao Family Comprehensive (Site 210), Orange, California
  - Karmanos Cancer Institute (Site 070), Detroit, Michigan